CLINICAL TRIAL: NCT03544476
Title: Interactive Mobile Health Intervention to Support Patients With Active Tuberculosis
Brief Title: Mobile Health Intervention for Active Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Sarah Iribarren, Assistant Professor, Biobehavioral Nursing and Health Informatics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00002080; K23NR017210 (NIH)
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Tuberculosis; Adherence, Medication
Keywords: mobile Health
MeSH Terms: conditions — Tuberculosis; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone TB treatment support app (Experimental): Daily use of the mobile phone TB treatment support app plus usual care. Participants will be asked to self-report daily TB medication administration, side-effects when applicable, and complete the direct adherence paper-based test randomly on 3-4 days of the week during the intensive treatment phase (first two months) and then 1-2 times per week during the maintenance phase (about month 3-6).
  Interventions: Behavioral: Mobile phone TB treatment support app plus usual care; Other: Usual care
- Usual care (Active Comparator): Usual care consists of outpatient treatment management from the time of diagnosis (unless symptoms are severe and hospitalization is recommended), routine clinical and laboratory tests, and follow-up appointments determined by the clinician. In general, patients receive 1-2 month's supply of medication and are asked to return monthly for follow-up.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Mobile phone TB treatment support app plus usual care — The behavioral intervention is delivered through a mobile phone TB support app. The functions allow the participant to: self-report daily administration of their TB medication, self-report side effects if applicable, review educational material on TB disease and its treatment, complete a treatment adherence monitoring test (urine drug metabolite test), take notes, and review their treatment progress/report. The drug metabolite test will require that the participant place a small amount of urine on the end of the paper strip, wait for results, and take a picture of the paper using the app. The purpose of this test is to confirm that medication was correctly taken within the past 24 hours.
  Arms: Mobile phone TB treatment support app
Other: Usual care — Usual care consists of outpatient treatment management from the time of diagnosis (unless symptoms are severe and hospitalization is recommended), routine clinical and laboratory tests, and follow-up appointments determined by the clinician. In general, patients receive 1-2 month's supply of medication and are asked to return monthly for follow-up.

SUMMARY:
The purpose of this study is to evaluate and further refine a mobile support tool for patients receiving treatment for active tuberculosis. Half of participants will receive support and monitoring using a mobile phone software application and usual care, while the other half will receive usual care.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a top ten leading cause of death globally despite it being a largely curable disease. New effective treatment supervision strategies are needed particularly in low-resource high TB burden settings and a potential solution is in the hands of nearly every patient - a mobile phone. Modern modular design mobile phone software applications ("apps") hold great promise to address this unmet need.

Current technologies allows for rapid design modification based on end user needs, implementation of native operating system (e.g., Android) versions for users with inconsistent internet access, and the integration of the patients' experiences with electronic health records using industry standards. Apps can perform multiple functions (e.g., automated reminders, symptom tracking, secure messaging, multi-media education). To date, few TB related apps have focused on patients as users, and none support patient engagement in self-management of their care or direct adherence monitoring. The research objectives are to understand end user needs and other stakeholder needs to build, refine, and pilot test an app to support patients self-administering treatment for active TB.

ELIGIBILITY:
Inclusion Criteria:

* Subject is starting TB treatment for the first time
* Subject has no known TB drug resistance
* Subject is HIV negative (self-reported or documented)
* Subject owns or has regular access to a mobile phone that can access the Internet and is able to operate the mobile phone to communicate or have someone able to assist.

Exclusion Criteria:

* Severely ill (i.e., requiring hospitalization)
* Reside in the same household with another study participant
* History of known drug resistance and HIV co-infection because their care is managed separately and the treatment regimens and duration differ.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Iribarren, PhD, RN, Principal Investigator — University of Washington
Locations (1):
- Hospital Dr. Antonio A. Cetrángolo, Vicente López, Province of Buenos Aires, Argentina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Phone TB Treatment Support App | Usual Care
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile Phone TB Treatment Support App | Usual Care | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 4 | 1 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (17.6) | 31.5 (14.3) | 36.5 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 10 | 11 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 21 | 42
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 17 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 4 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success
Description: Treatment outcomes will be measured using standard definitions set by the World Health Organization (WHO) Standards of TB treatment. Treatment success based on WHO definitions: completed (without bacteriological confirmation) or cured (negative sputum smear at 6 months and at least once prior to 6 months)). Other treatment outcomes include: failed (sputum smear positive at 5 months or later), died, defaulted (treatment interruption for ≥ 2 months), lost to follow-up (diagnosed, treatment outcome not documented), or transferred out (transferred to another reporting unit and treatment outcome is unknown).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Phone TB Treatment Support App | Usual Care
Number analyzed (Participants) | 21 | 21
Participants | 20 | 17

2. Secondary Outcome: Engagement: Average Number of Days Participants Reported Through the App
Description: Level of engagement using the app measured by the average number of days reporting treatment adherence over 180 days of treatment.
Time Frame: 6 months
Population: Intervention group only
Measure: Mean (Standard Deviation); unit: days reporting adherence
Arm/Group | Mobile Phone TB Treatment Support App | Usual Care
Number analyzed (Participants) | 21 | 0
days reporting adherence | 147.2 (34.4) |

3. Other Pre Specified Outcome: Feasibility of Implementation
Description: number of participants with access to a phone and internet connection
Time Frame: 6 months
Population: regular access to phone and internet connection
Measure: Count of Participants; unit: Participants
Arm/Group | Mobile Phone TB Treatment Support App | Usual Care
Number analyzed (Participants) | 20 | 21
Participants | 10 | 6

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Mobile Phone TB Treatment Support App | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/21 | 1/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03544476/Prot_SAP_000.pdf